CLINICAL TRIAL: NCT00804388
Title: Comparing Polyethylene Wear Using 3. Generation Highly Crosslinked Polyethylene in an Uncemented Total Hip Prostheses With Either 32 mm or 36 mm Caput of Ceramics
Brief Title: Wear Measurements of E-Poly in an Uncemented THA With Either 32 or 36 mm Caput of Ceramics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lovisenberg Diakonale Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government); Zimmer Biomet (Industry); Ullevaal University Hospital (Other)
Responsible Party: Einar Lindalen, MD, Lovisenberg Diakonale sykehus, Lovisenberg Diakonale sykehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-08366a; 03-2008 LDS
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Primary Arthrosis; Osteoarthritis
Keywords: Vitamine E; E-poly; Hip; Degenerative joint disease
MeSH Terms: conditions — Osteoarthritis; Joint Diseases | interventions — Arthroplasty, Replacement, Hip; Papaverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Uncemented total hip replacement, 32 mm caput
  Interventions: Procedure: Total hip arthroplasty
- 2 (Active Comparator): Uncemented total hip replacement, 36 mm caput
  Interventions: Procedure: Total hip arthroplasty

INTERVENTIONS:
Procedure: Total hip arthroplasty — 32 mm versus 36 mm caput of ceramics Vitamin E stabilized polyethylene
  Other Names: E-poly, Vitamine E, Hip, degenerative joint disease

SUMMARY:
The aim of the study is to compare polyethylene wear in an uncemented total hip prosthesis with 3rd. generation highly cross-linked polyethylene with a 32 mm ceramic femoral head compared to a 36 mm ceramic head. Using X-ray, RSA and DEXA.

The polyethylene to be used is E-Poly (Biomet).

The H0 hypothesis is that there is no difference with regard to polyethylene wear and bone loss between the two groups.

DETAILED DESCRIPTION:
Uncemented THA, 32 mm or 36 mm caput of ceramics, E-Poly inserts. Measure wear with RSA, X-Ray and bone mineral density with DEXA.

ELIGIBILITY:
Inclusion Criteria:

* 50-65 years old
* Primary or secondary osteoarthritis

Exclusion Criteria:

* Significant anatomical divergence are excluded
* Rheumatoid arthritis
* Fracture sequelae
* Dysplasia
* Immune suppression or grave systemic illness

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Measure polyethylene wear and bone mineral density between the two groups | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M. Røhrl, MD,PhD, Study Chair — Ullevål Univeristy Hospital Norway; Einar Lindalen, MD, Study Chair — Lovisenberg Diakonale sykehus
Locations (1):
- Lovisenberg Diakonale sykehus, Oslo, Norway